CLINICAL TRIAL: NCT01536340
Title: Identifying Adverse Events After Discharge From a Community Hospital
Status: Completed | Type: Observational
Sponsor: Florida State University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dennis Tsilimingras, MD, MPH, School of Medicine, Wayne State University
Other Study IDs: R01HS018694 (AHRQ)
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Iatrogenic Injury
Keywords: post discharge adverse events; discontinuities in care; medical injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to:

-Determine the incidence of adverse events, preventable adverse events, and ameliorable adverse events, and the timeliness of post-discharge ambulatory appointments, affecting urban and rural patients approximately 3-4 weeks after discharge from a hospitalist-run medical service of a large community hospital to home.

H1: The incidence of post-discharge adverse events will be higher in rural patients compared with urban patients discharged from a hospitalist-run medical service of a large community hospital.

-Identify and classify the types of post-discharge adverse events (e.g., adverse drug events, procedure-related events, hospital acquired (nosocomial) infections, falls, and other) affecting urban and rural patients approximately 3-4 weeks after discharge from a hospitalist-run medical service of a large community hospital to home.

H2: All patients will be at higher risk for adverse drug events than other types of adverse events.

-Examine the relationships between the population at risk, characteristics of the health care delivery system, and the utilization of post-discharge health services, and how these relationships help us understand the incidence of post-discharge adverse events.

H3: Several factors will be independently associated with the incidence of post-discharge adverse events in rural and urban patients, including patient comorbidity, severity of acute illness, presence of a primary care physician prior to hospitalization, and a scheduled timely post-discharge ambulatory follow-up appointment.

DETAILED DESCRIPTION:
This 24-month prospective cohort study will examine the frequency and types of adverse events experienced by patients 3-4 weeks after discharge from the Tallahassee Memorial Hospital (TMH), the timeliness of post-discharge ambulatory appointments, and identify the associations, if any, of readily available patient, system, and patient care factors with the occurrence of these post-discharge adverse events. Data collection will involve telephone interviews with patients, and review of inpatient and outpatient health records for services received, as necessary, within 3-4 weeks after discharge from the hospital. These data sources will allow study physicians to implicitly (with some explicit guidance) determine whether an adverse event has occurred, distinguish preventable from ameliorable adverse events, and determine the types of adverse events. In addition, the study will determine the timeliness of post-discharge ambulatory appointments by conducting post-discharge telephone interviews with patients and reviewing health records.

ELIGIBILITY:
Inclusion Criteria:

* age over 21 years
* discharged home from TMH general medical service
* patients must have a telephone number where they can be reached for an interview
* patient or surrogate must be able to interview in Spanish or English

Exclusion Criteria:

* age less than 21 years
* patient or surrogate non-English or Spanish speaking
* patients being discharged to an institutionalized care (assisted living facilities, prisons, etc.)
* patients not discharged from general medical service

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study population includes patients 21 and older living in Florida, who are discharged home from the TMH hospitalist service. Patients must have a phone number where they can be reached. They must also speak English or Spanish. Surrogates are permitted to complete an interview in the event that a patient is unable to complete it.
  Rural patients are those who live in counties where the population density is 100 people per square mile or less. Patients with diminished mental capacity are at increased risk of adverse events. These patients (or their surrogates) are included in the sample.
Sampling Method: Non-Probability Sample
Enrollment: 684 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
post discharge adverse event | six weeks after discharge from the hospital
  Patients are contacted 3-6 weeks after discharge for a phone interview. They are questioned about potential adverse events following their discharge from the hospital. Interviewers/nurses conduct a review of systems to determine if the patient experienced an adverse event. Potential cases are flagged on the basis of unexpected health care utilization, new/exacerbated symptoms and/or abnormal lab test results. Cases are reviewed by two independent physician reviewers to determine whether the adverse event was preventable, using their implicit judgment.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Tsilimingras, MD, MPH, Principal Investigator — Wayne State University; Ashley Duke, Study Director — Florida State University, College of Medicine
Locations (1):
- Tallahassee Memorial Healthcare, Tallahassee, Florida, United States

REFERENCES:
- [Background] Tsilimingras D, Schnipper J, Duke A, Agens J, Quintero S, Bellamy G, Janisse J, Helmkamp L, Bates DW. Post-Discharge Adverse Events Among Urban and Rural Patients of an Urban Community Hospital: A Prospective Cohort Study. J Gen Intern Med. 2015 Aug;30(8):1164-71. doi: 10.1007/s11606-015-3260-3. Epub 2015 Mar 31. PMID 25822112